CLINICAL TRIAL: NCT06657885
Title: Phase II, Pilot Study, Open Label, Multicenter, Evaluating Dual Antiretroviral Therapy With Long-acting Cabotegravir/Lenacapavir
Brief Title: CAbotégravir LENacapavir DUal Long Acting
Acronym: CALENDULA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No response regarding coverage of treatments by social security and the DGOS
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMEA 069; 2024-516028-33-01 (EU CTIS Number)
Record Dates: First submitted 2023-06-22; First posted 2024-10-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2024-09

CONDITIONS: HIV1 Infection; Multi-treated Patients Who Have Received Multiple Lines of Antiretroviral Treatment; CABOTEGRAVIR; LENACAPAVIR; Stable Oral Antiretroviral Treatment for at Least 6 Months
Keywords: CAbotégravir LENacapavir DUal Long Acting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm (Experimental)
  Interventions: Drug: his is a prospective, single-arm, multicentre, non-randomised phase II, pilot study designed to achieve or maintain virological success in participants who meet the prescribing criteria for lenacapavi

INTERVENTIONS:
Drug: his is a prospective, single-arm, multicentre, non-randomised phase II, pilot study designed to achieve or maintain virological success in participants who meet the prescribing criteria for lenacapavi — cabotegravir initiation: daily oral route of 1 tablet 30 mg at Day 0 to week 4 Cabotegravir maintennace: Every 8 weeks (+/- 1 week) intramuscular injection from week 8 at week 48.
  Lenacapavir initiation: Subcutaneous injection (927mg/3ml),ie 2 injections of 463,5mg/1,5mL in 2 distinct abdominal sites + orale route of 2 tablets of 300mg (ie 600 mg) at Day 0 and at day 1: orale route of 2 tablets of 300mg (ie 600 mg) Lenacapavir maintenance: Subcutaneous injection (927mg/3ml),ie 2 injections of 463,5mg/1,5mL in 2 distinct abdominal sites every 24 weeks (+/-1 week) from Day 0 to Week 48

SUMMARY:
This study is a Phase II, prospective, single-arm, multicenter, non-randomized pilot study designed to evaluate the antiretroviral efficacy of lenacapavir in combination with cabotegravir injection over 48 weeks of follow-up in participants who meet the study inclusion criteria. Efficacy is defined as the absence of virologic failure at S48. Virologic success is defined as maintaining or achieving CV < 50 copies/mL without interruption of long-acting dual therapy with cabotegravir/lenacapavir at the end of 48 weeks. The study will be conducted at several sites in France in adults 18 years of age and older. Minors and persons under legal guardianship will not be included in the study.

Long-acting treatments are evolving thanks to new "long-acting" molecules. These molecules ensure prolonged efficacy without the need for daily dosing thanks to their long half-life by oral / IM or SC injection (cabotegravir, islatravir, lenacapavir, rilpivirine and bNAbs).

Currently, the only available combination is dual therapy with cabotegravir/rilpivirine administered intramuscularly every two months. However, this injectable combination therapy has its limitations, namely previous resistance to rilpivirine, a number of failures due to certain virological subtypes or poor use of the injectable by certain patients (obesity, injection errors, etc.). For many referral centers caring for patients with HIV, it has become necessary to have a long-acting therapeutic alternative for certain patients. A strategy based on lenacapavir combined with cabotegravir could be a validated alternative for undetectable or detectable patients who have received intensive multidrug regimens, for patients with multidrug resistance, or for patients who are unable to take their oral antiretroviral regimens due to intolerance, drug-drug interactions, or non-adherence.

Recently in the US, the case series presented by Dr. Monica Gandhi (Case series examining the Long-Acting combination of Lenacapavir and Cabotegravir: call for a trial-abstract 629 CROI 2024) demonstrated the high virologic efficacy (94%) of this combination in participants who were unobserved, intolerant or had underlying resistance to antiretroviral therapy (NNRTIs).

The experimental drugs used in this study are cabotegravir, marketed as Vocabria®, and lenacapavir, marketed as Sunlenca®. Both are approved in France for the treatment of HIV-1 infection.

ELIGIBILITY:
Age ≥ 18 years

* HIV-1 infection
* Stable oral antiretroviral treatment for at least 6 months
* Multi-treated patients who have received multiple lines of antiretroviral treatment
* Undetectable patients with CV < 50 copies/mL in the last 6 months (a single blip between 50 and 200 copies/mL in the last 6 months is allowed) and eligible to switch to the lenacapavir/cabotegravir strategy on the basis of a collegial decision by clinicians, virologists and pharmacologists following a multidisciplinary meeting due to
* the presence of resistance mutations, including to NNRTIs
* or oral drug intolerance
* or drug-drug interactions
* Detectable, virologically uncontrolled HIV viral load ≥ 200 c/mL in the last 12 months who is eligible to switch to the lenacapavir/cabotegravir strategy based on a collegial decision by clinicians, virologists and pharmacologists following a multidisciplinary meeting due to
* the presence of resistance mutations, including to NNRTIs
* or oral drug intolerance
* or drug-drug interactions
* ASAT and ALAT < 3N
* Creatinine GFR > 60 mL/min (CKD-EPI)
* Haemoglobin > 10 g/dL
* Platelets > 100 000/mm3
* Commitment to use preventive and protective means of sexual intercourse for the duration of the trial.
* For women at risk of pregnancy, commitment to use an effective method of contraception for the duration of the study.
* Affiliated or beneficiary of a social security scheme (article L1121-11 of the French Public Health Code),
* Free, informed, written consent, signed by the person and the investigator no later than the day of inclusion and before any examination carried out as part of the study (article L1122-1-1 of the French Public Health Code).

Non-inclusion criteria

* HIV-2 infection or HIV-1/HIV2 co-infection
* HIV-1 subtype A6/A1
* BMI ≥ 30kg/m².
* Chronic active viral hepatitis B with positive Hbs antigen
* Active chronic viral hepatitis C requiring specific treatment over the next 48 weeks.
* Treatment with interferon, interleukin or any other immunotherapy or chemotherapy in progress.
* Active opportunistic infection, or acute treatment for opportunistic infection
* Any condition (alcohol, drugs, neurological or neuropsychiatric disorders, etc.) likely to compromise tolerance of treatment and/or patient compliance with treatment and adherence to the protocol, as judged by the investigator.
* Women who are breastfeeding, pregnant or refusing contraception
* Taking medication contraindicated with the trial treatment
* Major incapacity, legal protection, guardianship or curatorship
* Planning to move house within the next 18 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with virological failure | week 48
Percentage of participants with virological failure | Week 24

SECONDARY OUTCOMES:
Percentage of participants with virological failure | Week 24, week48
Percentage of participants achieving therapeutic success at W48 (absence of virological failure and definitive discontinuation of assigned treatment or study continuation due to intolerance). Change of residence, change of treatment due to pregnancy, for | week 48
Percentage of participants with viruses harbouring resistance mutations to the current treatment at the time of virological failure (by Sanger) and description of the resistance mutations selected at the time of virological failure. | at the time of virologic failure
Proportion of minority resistance variants archived in DNA at D0 and their impact on the risk of virological failure and on the selection of resistance mutations. | D0
Describe the evolution of the proportion of intact and defective proviruses in PBMC at D0 and W48. | day 0 and week 48
Percentage of participants with at least one "blip" (viral load greater than 50 copies/mL with a control less than or equal to 50 copies/mL) between D0 and W48. | Between day 0 and week 48
Change in CD4 and CD8 T lymphocytes and CD4/CD8 ratio between W-2 and W48 | Week -2 and week 48
Description of plasma concentrations of antiretroviral treatments between D0 and W48 | between day0 and week 48
Incidence of clinical and laboratory grade 3 or higher adverse events | betwwen Day 0 and week 48
Incidence of adverse events and discontinuation from study to W48 | Between day 0 and week 48
Changes in weight and BMI from D0 to W48 | Between day 0 and week 48
Metabolic parameters (total cholesterol, LDL-c, HDL-c, triglycerides and fasting plasma glucose) from D0 to W48 | Between day 0 and week 48
Change in participants' symptoms as assessed by self-report questionnaire from D0 to W48 | Between day 0 and week 48
Assessment of participant satisfaction by questionnaire between D0 and W48 | Between day 0 and week 48
Percentage of participants with virological failure | week24 and week 48
Percentage of participants with virological failure | week24

CONTACTS AND LOCATIONS:
Overall Officials: Roland LANDMAN, Principal Investigator — IMEA and Bichat hospital
Locations (12):
- France (12):
  - Hopital Saint André, Bordeaux
  - Hopiytal Pellegrin, Bordeaux
  - Centre hospitalier François Mitterrand, Dijon
  - Hopital raymond Poincaré, Garches
  - Hôpital Franco-Britannique, Levallois-Perret
  - CHU de nantes- Hotel Dieu, Nantes
  - Chu- Nice Archet, Nice
  - Hopital Saint Antoine, Paris
  - Hopital Pitié Salpêtrière, Paris
  - Hopital Necker, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Centre hospitalier de Tourcoing, Tourcoing

IPD SHARING:
Plan to Share IPD: Undecided